CLINICAL TRIAL: NCT02882191
Title: Evaluation of the Effectiveness, Safety and Tolerability of LevoCept (Levonorgestrel-Releasing Intrauterine System) for Long-Acting Reversible Contraception
Brief Title: Evaluation of the Efficacy and Safety of LevoCept
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sebela Women's Health Inc. (Industry)
Collaborators: Synteract, Inc. (Industry)
Responsible Party: Sponsor
Organization: Sebela Pharmaceuticals Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMDOC-0022
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Contraception
Keywords: contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LevoCept IUD (Experimental): LevoCept IUD placement
  Interventions: Drug: LevoCept

INTERVENTIONS:
Drug: LevoCept — placement of LevoCept IUD
  Other Names: Levonorgestrel-Releasing Intrauterine System

SUMMARY:
To evaluate the effectiveness, device placement, safety, and tolerability of LevoCept to support commencing a Phase III Clinical Study

DETAILED DESCRIPTION:
Study Design:

Prospective, multi-center, single-arm, open-label, Phase II clinical study

Approximately 250 subjects will be enrolled at about 14 centers in the US.

Study Population: Pre-menopausal women ages 18 - 40, at risk for pregnancy, who are interested in using only this intrauterine contraceptive for birth control will be eligible for this study. Subjects must provide written informed consent and meet the study subject selection criteria without any exclusions as outlined in the Clinical Investigation Plan (CIP).

Primary Effectiveness Outcome:

The primary outcome measure is effectiveness, evaluated as the absence of pregnancy during LevoCept use.

Safety and other outcome measures include:

Study Device Placement:

* Ease of placement
* Placement success

Safety:

* Serious Adverse Events
* Adverse Events

Tolerability:

* Bleeding and spotting patterns
* Discontinuation rate and reasons for discontinuation

ELIGIBILITY:
Inclusion Criteria:

1. Between 18-40 years of age at the time of study initiation; 1.1 Enrollment will be targeted for 225 subjects aged 18-35 (for safety and effectiveness analyses) and an additional 25 subjects aged 36-40 (for safety only) (note: all subjects will be included in the analysis for device placement and tolerability);
2. Pre-menopausal, as determined by regular menstrual cycle (28 ± 7 days) for the last 3 months; 2.1 Based on patient history, when not on hormonal contraceptives;
3. Sexually active with a male partner who has not had a vasectomy;
4. Reasonably expected to have to coitus at least once monthly during the study period.
5. In a mutually monogamous relationship of at least 3-6 months duration;
6. Seeking to avoid pregnancy for the next 12 months;
7. Willing to use the study device as the sole form of contraception;
8. Willing to accept a risk of pregnancy;
9. Normal PAP or ASC-US with negative high risk HPV test result within the appropriate screen timeframe, and prior to LevoCept insertion;
10. Able and willing to comply with all study tests, procedures, assessment tools and follow-up; and
11. Able and willing to provide and document informed consent and Authorization for Release of Protected Health Information (PHI).

Exclusion Criteria:

1. Known or suspected pregnancy; or at risk for pregnancy from unprotected intercourse earlier in current cycle
2. Subject who anticipates separation from her partner for more than 1 cycle within the next 12 months;
3. A previously inserted IUD that has not been removed by the time LevoCept is placed;
4. History of previous IUD complications, such as perforation, expulsion, infection (pelvic inflammatory disease) or pregnancy with IUD in place.;
5. Injection of hormonal contraceptive (e.g., Depo-Provera) within the last 10 months; 5.1 Must have had 2 normal menstrual cycles since the last injection;
6. Planned use of any non-contraceptive estrogen, progesterone or testosterone any time during the 12 months of study participation;
7. Postpartum, prior to a minimum of 6 weeks and complete uterine involution;
8. Exclusively breastfeeding before return of menses; Lactating women will be excluded unless they have had have had two normal menstrual periods prior to enrollment.

   8.1 Must have had 2 normal spontaneous menstrual cycles since delivery
9. Unexplained abnormal uterine bleeding (suspicious for serious condition), before evaluation; Immediately post-septic abortion or puerperal sepsis;
10. Severely heavy or painful menstrual bleeding;
11. Suspected or known cervical, uterine or ovarian cancer, or unresolved clinically significant abnormal pap smear requiring evaluation or treatment.
12. Any history of gestational trophoblastic disease with or without detectable elevated ß-hCG levels, or related malignant disease without an intervening normal pregnancy;
13. Any congenital or acquired uterine anomaly that may complicate IUD placement, such as:

    13.1 Submucosal uterine leiomyoma 13.2 Asherman's syndrome 13.3 Pedunculated polyps 13.4 Bicornuate uterus 13.5 Didelphus or uterine septa
14. Any distortions of the uterine cavity (e.g. fibroids), in the opinion of the investigator, likely to cause issues during insertion, retention or removal of the IUD;
15. Known anatomical abnormalities of the cervix such as severe cervical stenosis, prior trachelectomy or extensive conization that, in the opinion of the investigator would prevent cervical dilation and study device placement;
16. Current or recent (within the last 3 months) untreated acute cervicitis or vaginitis;
17. Known or suspected breast cancer or other progestin-sensitive cancer now or in the past;
18. Known acute liver disease or liver tumor;
19. Subjects who have an established immunodeficiency;
20. High risk for STDs (e.g., multiple sexual partners);
21. Known or suspected HIV infection or clinical AIDS;
22. Known intolerance or allergy to any component of the LevoCept system; including nickel, silicone or tantalum;
23. Subject had LevoCept placed previously or had 2 attempts at placement;
24. Known or suspected alcohol or drug abuse within 12 months prior to the screening visit;
25. Any general health or behavioral condition that, in the opinion of the Investigator, could represent an increased risk for the subject or would render the subject less likely to provide the needed study information.
26. Subject is currently participating or has participated in another clinical study involving another investigational agent within 30 days of the planned LevoCept insertion date or is planning participation in another clinical trial with an investigational agent within 52 weeks (visit 6) after insertion.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 279 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
absence of pregnancy during LevoCept use | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David Turok, MD, Principal Investigator — University of Utah
Locations (16):
- United States (16):
  - Essential Access Health-Berkeley, Berkeley, California
  - Essential Access Health-Los Angeles, Los Angeles, California
  - University of California Davis Health System Department of Obstetrics and Gynecology, Sacramento, California
  - University Of Colorado Department of Obstetrics & Gyncology, Aurora, Colorado
  - Healthcare Clinical Data, Inc., North Miami, Florida
  - Emory University School of Medicine Gynecology/Obstetrics, Atlanta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Columbia University Medical Center, New York, New York
  - University of Cincinnati Physicians Company, Inc, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Clinical Research of Philadelphia, LLC, Philadelphia, Pennsylvania
  - Advanced Research Associates, Corpus Christi, Texas
  - University of Utah Healthcare Health Sciences Center, Salt Lake City, Utah
  - Seattle Women's: Health, Research, Gynecology, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No